CLINICAL TRIAL: NCT03803150
Title: A Comparative Study Between Preauricular Retromandibular Anteroparotid Approach and Retromandibular Transparotid Approach in Internal Fixation of Subcondylar Fracture on Facial Nerve Injury and Parotid Fistula
Brief Title: Evaluation of Preauricular Retromandibular Anteroparotid Versus Retromandibular Through Parotid Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Hani Taher Hibatullah Ali, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TMAP in subcondylar fracture
Record Dates: First submitted 2018-12-24; First posted 2019-01-14 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Subcondylar Process of Mandible Open Fracture; Facial Nerve Injuries
MeSH Terms: conditions — Facial Nerve Injuries

STUDY DESIGN:
Intervention Model Description: Block, consecutive, 1:1 Consecutive because patients with subcondylar fracture need immediate surgical intervention, that is why investigators can not wait to collect the whole sample size and make computer generated randomization .
Masking Description: Senior supervisor Prof. Dr. Hairy El mossy will generate the allocation sequence.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRA approach (Experimental): PRA extends downward in curvilinear fashion in cervicomastoid skin crease
  Interventions: Procedure: PRA approach
- RT approach (Active Comparator): RT begins 5mm below the ear lobe and continues 3 to 3.5cm inferiorly.
  Interventions: Procedure: RT approach

INTERVENTIONS:
Procedure: PRA approach — A preauricular incision will be made that extends downwards in a curvilinear fashion in the cervicomastoid skin crease, though any variation in this incision will suffice. The great auricular nerve will be preserved and the flap raised in the subdermal fat plane, superficial to the superficial musculoaponeurotic layer to allow access to the masseter adjacent to the anteroinferior edge of the parotid gland, just below the parotid duct. Branches of the facial nerve will be readily identified and avoided with or without loupe magnification, on the surface of the masseter muscle.
  Arms: PRA approach
Procedure: RT approach — The incision for the retromandibular approach begins 5mm below ear lobe and continues 3 to 3.5cm inferiorly. Initial incision begins through skin and subcutaneous tissues,platysma muscle ,(SMAS), parotid capsule Dissection is continued until the only tissue remaining on the posterior border of the mandible will be the periosteum of pterygomassetric sling,then the fracture site will exposed and reduced.
  Arms: RT approach

SUMMARY:
Of all the bones in the maxillofacial area, the condylar process is the most susceptible to fracture. The incidence of condylar fracture accounts for 25% to 50% of all mandibular fractures. Though remained controversial for a long time, surgical treatment of displaced subcondylar fractures appears today as the gold standard.

Although there is a developing preference for open reduction and internal fixation of mandibular condylar fractures, the optimal approach to the ramus condylar unit remains controversial. Various approaches have been proposed, and each has specific shortcomings and disadvantages. Retromandibular, submandibular, transoral, and through parotid approaches are generally performed and sometimes used with an endoscope. Limited access and injury to the facial nerve are the most common problems, while Wilson introduced a new through masseter anteroparotid approach, this technique offers excellent access to the ramus condylar unit, and facial nerve damage risk is reduced.

DETAILED DESCRIPTION:
Fractures of the mandibular condylar process have been documented to be one of the most common occurring mandibular fractures.

When open treatment is selected, several surgical approaches can be used to expose, reduce, and stabilize the fracture site, each with its own set of advantages and disadvantages. Surgical approaches to the fractured mandibular condyle are broadly classified into intraoral and extraoral approaches. Intraoral approaches can be performed with or without endoscopic assistance. The most common extraoral approaches are submandibular, Risdon, preauricular, retroauricular, and retromandibular through parotid or through masseter approaches.

An intraoral approach is time consuming and requires special instruments such as an endoscope, and additional training. Furthermore, cases of high fractures and/or medially displaced condylar fractures are technically difficult to manage through an intraoral approach, incorrect anatomical reduction, condylar head resorption, myofascial pain, and malocclusions have been reported to be more common complications following the intraoral approach when compared to extraoral approaches.

In contrast, extraoral approaches are commonly used because they produce better visualization of the fracture site and therefore facilitate fracture reduction and fixation. However, extraoral approaches are complicated by the risk of injury to the facial, great auricular, and auriculotemporal nerves, visible scars, sialoceles, Frey syndrome and salivary fistulas.

ELIGIBILITY:
Inclusion Criteria:

1. Patients age should be more than 18 year.
2. Patients with subcondylar fracture and need to open reduction and internal fixation using titanium miniplates.
3. Patients should be free from any traumatic injuries to facial nerve or parotid gland.
4. Availability of preoperative and postoperative panoramic radiographs and/or computed tomography (CT) images.
5. Mental status permitting an adequate neuromotor examination.
6. Regular clinical follow-up, documented in our clinical and radiographic evaluation charts, at 1 week, 1 month, 3 months and 6 months postoperatively

Exclusion Criteria:

1. Intraoral treatment of subcondylar fracture.
2. Incooperative patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-05-08 (Actual)

PRIMARY OUTCOMES:
Minimize facial nerve injury | Concerning the facial injury will be at 6 months
  Regarding facial nerve injury the measuring device is House- brachmann facial nerve grading system (HBFNGS) while the measuring unit is numerical from (I-VI) I= Normal, II= Mild dysfunction, III= Moderate dysfunction, IV= Moderately severe dysfunction, V= Severe dysfunction, VI= Total paralysis.
  I= Better while VI= Worse
Minimize salivary fistula | Salivary fistula at 1 week
  Regarding salivary fistula the measuring device is clinical examination while the measuring unit is binary question.

SECONDARY OUTCOMES:
Reduce scar formation | at 6 months
  The character of any observed scar was scored as (1) no perceptible scar, (2) visible but thin and linear scar, (3) wide scar, and (4) hypertrophic scar or keloid. while the measuring unit is numerical from (1-4)
  1= Better while 4= Worse

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dental and oral medicine / Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Once I finished the study I will share the data

REFERENCES:
- [Result] Tang W, Gao C, Long J, Lin Y, Wang H, Liu L, Tian W. Application of modified retromandibular approach indirectly from the anterior edge of the parotid gland in the surgical treatment of condylar fracture. J Oral Maxillofac Surg. 2009 Mar;67(3):552-8. doi: 10.1016/j.joms.2008.06.066. PMID 19231779
- [Result] Lutz JC, Clavert P, Wolfram-Gabel R, Wilk A, Kahn JL. Is the high submandibular transmasseteric approach to the mandibular condyle safe for the inferior buccal branch? Surg Radiol Anat. 2010 Dec;32(10):963-9. doi: 10.1007/s00276-010-0663-z. Epub 2010 May 12. PMID 20461515
- [Result] Guerrissi JO. A transparotid transcutaneous approach for internal rigid fixation in condylar fractures. J Craniofac Surg. 2002 Jul;13(4):568-71. doi: 10.1097/00001665-200207000-00018. PMID 12140424
- [Result] Ozkan HS, Sahin B, Gorgu M, Melikoglu C. Results of transmasseteric anteroparotid approach for mandibular condylar fractures. J Craniofac Surg. 2010 Nov;21(6):1882-3. doi: 10.1097/SCS.0b013e3181f4aef7. PMID 21119445
- [Result] Wilson AW, Ethunandan M, Brennan PA. Transmasseteric antero-parotid approach for open reduction and internal fixation of condylar fractures. Br J Oral Maxillofac Surg. 2005 Feb;43(1):57-60. doi: 10.1016/j.bjoms.2004.09.011. PMID 15620776
- [Result] Zachariades N, Papavassiliou D. The pattern and aetiology of maxillofacial injuries in Greece. A retrospective study of 25 years and a comparison with other countries. J Craniomaxillofac Surg. 1990 Aug;18(6):251-4. doi: 10.1016/s1010-5182(05)80425-1. PMID 2212022
- [Result] Villarreal PM, Monje F, Junquera LM, Mateo J, Morillo AJ, Gonzalez C. Mandibular condyle fractures: determinants of treatment and outcome. J Oral Maxillofac Surg. 2004 Feb;62(2):155-63. doi: 10.1016/j.joms.2003.08.010. PMID 14762747
- [Result] Choi BH, Yoo JH. Open reduction of condylar neck fractures with exposure of the facial nerve. Oral Surg Oral Med Oral Pathol Oral Radiol Endod. 1999 Sep;88(3):292-6. doi: 10.1016/s1079-2104(99)70030-2. PMID 10503856
- [Result] Salgarelli AC, Anesi A, Bellini P, Pollastri G, Tanza D, Barberini S, Chiarini L. How to improve retromandibular transmasseteric anteroparotid approach for mandibular condylar fractures: our clinical experience. Int J Oral Maxillofac Surg. 2013 Apr;42(4):464-9. doi: 10.1016/j.ijom.2012.12.012. Epub 2013 Feb 8. PMID 23395651
- [Result] Jensen T, Jensen J, Norholt SE, Dahl M, Lenk-Hansen L, Svensson P. Open reduction and rigid internal fixation of mandibular condylar fractures by an intraoral approach: a long-term follow-up study of 15 patients. J Oral Maxillofac Surg. 2006 Dec;64(12):1771-9. doi: 10.1016/j.joms.2005.12.069. PMID 17113444
- [Result] Schmidseder R, Scheunemann H. Nerve injury in fractures of the condylar neck. J Maxillofac Surg. 1977 Sep;5(3):186-90. doi: 10.1016/s0301-0503(77)80103-3. PMID 269890
- [Result] Weinberg S, Kryshtalskyj B. Facial nerve function following temporomandibular joint surgery using the preauricular approach. J Oral Maxillofac Surg. 1992 Oct;50(10):1048-51. doi: 10.1016/0278-2391(92)90488-l. PMID 1527657
- [Result] Handschel J, Ruggeberg T, Depprich R, Schwarz F, Meyer U, Kubler NR, Naujoks C. Comparison of various approaches for the treatment of fractures of the mandibular condylar process. J Craniomaxillofac Surg. 2012 Dec;40(8):e397-401. doi: 10.1016/j.jcms.2012.02.012. Epub 2012 Mar 21. PMID 22440318